CLINICAL TRIAL: NCT01289548
Title: Effect of Lower Limb Ischaemic Preconditioning on Renal Function in Patients Undergoing Living Donor Kidney Transplantation
Brief Title: Effect of Remote Ischaemic Preconditioning on Renal Function in Patients Undergoing Living Donor Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: B. Braun Medical SA (Industry)
Responsible Party: Principal Investigator, Hua Zheng, M.D. Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TJMZK201001
Record Dates: First submitted 2011-02-02; First posted 2011-02-03 (Estimated); Results first posted 2013-09-10 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Kidney Diseases; Kidney Failure, Chronic; Kidney Failure; Renal Insufficiency; Renal Insufficiency, Chronic; Urologic Diseases
Keywords: remote ischaemic preconditioning; kidney transplantation
MeSH Terms: conditions — Kidney Diseases; Kidney Failure, Chronic; Renal Insufficiency; Renal Insufficiency, Chronic; Urologic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (No Intervention): patients (both donors and recipients) had a deflated cuff placed on the left lower limb for 30 min
- donor (Experimental): Donors receive remote ischaemic preconditioning after anaesthesia induction and before surgery started; recipients only have a deflated blood pressure cuff around their leg for 30 minutes.
  Interventions: Device: remote ischaemic preconditioning
- recipient (Experimental): recipients receive remote ischaemic preconditioning after anaesthesia induction and before surgery started; donors only have a deflated blood pressure cuff around their leg for 30 minutes.
  Interventions: Device: remote ischaemic preconditioning

INTERVENTIONS:
Device: remote ischaemic preconditioning — Remote ischaemic preconditioning consisted of three 5-min cycles of left lower limb ischaemia, which was induced by an automated cuff-inflator placed on the left lower limb and inflated to 300 mm Hg, with an intervening 5 min of reperfusion during which the cuff was deflated.
  Other Names: RIPC
  Arms: donor; recipient

SUMMARY:
The purpose of this study was to investigate whether lower limb ischaemic preconditioning can improve renal function in patients undergoing living donor kidney transplantation

DETAILED DESCRIPTION:
Ischemia reperfusion injury (IRI) induced renal failure after kidney transplantation is a common clinical problem associated with a high morbidity and mortality. To reduce the adverse effects of IRI after organ transplantation various strategies aimed at the different pathophysiological processes of IRI have been investigated. Remote ischemic preconditioning (RIPC) is one such strategy where brief IRI of one organ protects other organs from sustained IRI. Many studies have shown that RIPC protects heart, muscle flaps, stomach, liver, lungs, and kidneys from IRI. RIPC of the limb with a tourniquet is a safe and convenient method of preconditioning organs against IRI. However, the efficacy of RIPC in patients undergoing living donor kidney transplantation need to be established and mechanism of early and late RIPC, such as whether the donor should undergo remote preconditioning or the recipient, need to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Subject capable of giving written informed consent, with end-stage kidney disease, who is a suitable candidate for primary kidney transplantation
* Living donors
* Compatible ABO blood type
* PRA < 20%

Exclusion Criteria:

* Re-transplant patients
* Those with peripheral vascular disease affecting the lower limbs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-05; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuke Tian, M.D., Study Chair — Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Department of Anaesthesiology, Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Chen Y, Zheng H, Wang X, Zhou Z, Luo A, Tian Y. Remote ischemic preconditioning fails to improve early renal function of patients undergoing living-donor renal transplantation: a randomized controlled trial. Transplantation. 2013 Jan 27;95(2):e4-6. doi: 10.1097/TP.0b013e3182782f3a. No abstract available. PMID 23325011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients scheduled for living donor renal transplantation in the Department of Transplantation, Tongji Hospital, Huazhong University of Science and Technology were recruited in the project from May 2010 to November 2011.
Pre-assignment Details: 68 pairs of patients were enrolled during the recruitment period. among them, 5 recipients had the history of renal transplantation before; 2 recipients had concomitant diabetes mellitus; and another one recipient had severe varicose vein in his lower limb. The left 60 pairs of donors and recipients (120 in total) were finally assigned to groups.
Groups:
- Donor RIPC: Donors receive remote ischaemic preconditioning after anaesthesia induction and before surgery started; recipients only have a deflated blood pressure cuff around their leg for 30 minutes.
- Recipient PIPC: recipients receive remote ischaemic preconditioning after anaesthesia induction and before surgery started; donors only have a deflated blood pressure cuff around their leg for 30 minutes.
Period: Overall Study
Arm/Group | Control | Donor RIPC | Recipient PIPC
Started | 40 (include both donors and recipients listed as milestones below) | 40 (include both donors and recipients listed as milestones below) | 40 (include both donors and recipients listed as milestones below)
Donors | 20 | 20 | 20
Recipients | 20 | 20 | 20
Completed | 40 | 40 | 40
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Donor + RIPC: Donors receive remote ischaemic preconditioning after anaesthesia induction and before surgery started; recipients only have a deflated blood pressure cuff around their leg for 30 minutes.
- Recipient +RIPC: recipients receive remote ischaemic preconditioning after anaesthesia induction and before surgery started; donors only have a deflated blood pressure cuff around their leg for 30 minutes.
- Total: Total of all reporting groups
Arm/Group | Control | Donor + RIPC | Recipient +RIPC | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age Continuous [Mean (Standard Deviation); unit: years] — Age of the recipient
  years | 32.5 (10.3) | 28.1 (6.5) | 30.6 (7.0) | 30.4 (8.2)
Age Continuous [Mean (Standard Deviation); unit: years] — Age of the donor
  years | 46.9 (6.4) | 47.4 (10.0) | 48.7 (5.2) | 47.6 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of the recipient
  Participants
    Female | 4 | 4 | 6 | 14
    Male | 16 | 16 | 14 | 46
Sex: Female, Male [Count of Participants; unit: Participants] — Gender of the donor
  Participants
    Female | 12 | 14 | 10 | 36
    Male | 8 | 6 | 10 | 24
Region of Enrollment [Number; unit: donors/recipients pairs]
  China | 20 | 20 | 20 | 60
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI of the recipient. BMI=weight(kg)/〖height(m)〗^2
  kg/m^2 | 20.08 (2.75) | 19.94 (1.99) | 20.38 (3.20) | 20.13 (2.65)
Cold ischemic time [Mean (Standard Deviation); unit: minutes] — Time from fully perfusion of the donor kidney to complement of the artery unclamping in the transplantation surgery
  minutes | 175.65 (36.35) | 166.25 (19.22) | 177.25 (27.59) | 173.05 (28.52)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI of the donor. BMI=weight(kg)/〖height(m)〗^2
  kg/m^2 | 22.19 (3.51) | 22.19 (2.43) | 23.45 (2.61) | 22.61 (2.90)
Relationship [Number; unit: donors/recipients pairs] — The donor's relationship with the recipient
  donors/recipients pairs
    parents | 12 | 16 | 14 | 42
    siblings | 6 | 2 | 5 | 13
    spouses | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Plasma Creatine Concentration of the Recipients
Description: Plasma creatinine concentration before surgery, 1hour, 4hours, 24hours, 48hours and 72hours after the artery unclamping
Time Frame: within the first 3days after the operation
Population: All patients completed the trial and no dropout occured.
Measure: Median (Inter-Quartile Range); unit: μmol/l
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
μmol/l
  before operation | 849.5 (122.34) [711.5 to 936.0] | 878.5 (258.41) [717.8 to 1143.5] | 771.0 (205.40) [559.5 to 860.3]
  1hour after the artery unclamping | 776.5 (102.74) [686.5 to 867.5] | 797.5 (231.99) [645.0 to 1060.0] | 725.5 (182.56) [636.8 to 814.5]
  4hours after the artery unclamping | 651.5 (118.27) [555.5 to 710.5] | 639.0 (226.72) [494.8 to 883.3] | 600.5 (213.39) [420.3 to 728.5]
  24hours after the artery unclamping | 222.5 (102.44) [183.5 to 329.5] | 240.5 (92.51) [166.5 to 353.0] | 253.5 (121.40) [163.0 to 382.0]
  48hours after the artery unclamping | 150.0 (80.35) [129.8 to 241.8] | 193.5 (74.69) [121.8 to 252.8] | 176.5 (96.18) [112.8 to 282.8]
  72hours after the artery unclamping | 120 (48.25) [110.5 to 167.0] | 153.0 (73.61) [98.8 to 216.3] | 126.5 (71.78) [98.5 to 225.3]

2. Secondary Outcome: Acute Rejection of Transplanted Kidney
Description: biopsy-confirmed, clinically symptomatic
Time Frame: before discharge
Population: All the patients completed the study and no dropout occured.
Measure: Number; unit: participants
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
participants | 0 | 0 | 0

3. Secondary Outcome: Delayed Graft Function
Description: Delayed Graft Function according to the clinical symptoms
Time Frame: before discharge
Population: All the patients completed the study and no dropout occured.
Measure: Number; unit: participants
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
participants | 1 | 2 | 2

4. Secondary Outcome: Length of Postoperative Hospital Stay
Description: time from the day of operation to the day of discharge for the recipients
Time Frame: before discharge
Population: All the patients completed the study and no dropout occured.
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
day | 17 (4.8) [15 to 21.8] | 15 (3.7) [14 to 16.8] | 14.5 (8.2) [13 to 24]

5. Primary Outcome: Urinary Output of the Recipients Postoperatively
Description: Accumulated urinary output 1hour, 4hours and 24hours after the artery unclamping and the urinary output on the 2nd and 3rd day after the operation
Time Frame: within the first 3days after the operation
Population: All patients completed the trial and no dropout occured.
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
ml
  within 1hour after the artery unclamping | 175 (265.1) [63 to 400] | 300 (239.6) [100 to 575] | 100 (220.4) [63 to 300]
  within 4hours after the artery unclamping | 1875 (1502.7) [1030 to 3338] | 2650 (1271.9) [1613 to 3600] | 1850 (999.8) [1138 to 2775]
  within 24hours after the artery unclamping | 8775 (5289.8) [5030 to 12588] | 10025 (5151.0) [4338 to 13850] | 6375 (3497.0) [4413 to 8888]
  on the 2nd day after the operation | 5355 (2051.7) [3838 to 7000] | 5200 (3846.3) [2900 to 6778] | 4020 (1984.5) [3438 to 5625]
  on the 3rd day after the operation | 4600 (1215.9) [3050 to 5348] | 3765 (2166.7) [2613 to 5138] | 3650 (1451.5) [2913 to 5260]

6. Primary Outcome: Plasma Concentration of NGAL in the Recipients
Description: Plasma concentration of neutrophil gelatinase-associated lipocalin (NGAL) before the operation and 24hours after the artery unclamping
Time Frame: within the first 24hours after the operation
Population: All patients completed the trial and no dropout occured.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
ng/ml
  before operation | 1478.7 (617.65) [976.1 to 1794.3] | 1269.1 (603.10) [1077.9 to 1839.2] | 1377.9 (677.98) [940.6 to 1838.5]
  24hours after the artery unclamping | 317.8 (210.41) [225.0 to 440.1] | 370.1 (212.51) [113.8 to 523.5] | 256.2 (309.04) [128.8 to 571.5]

7. Secondary Outcome: Total Costs During the Hospitalization
Description: Total costs from the admission to the discharge of the recipients
Time Frame: from the admission to the discharge of the patients
Population: All the patients completed the study and no dropout occured.
Measure: Median (Inter-Quartile Range); unit: RMB yuan
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
RMB yuan | 82499 (23625.18) [77320 to 127140] | 83574 (22164.70) [73912 to 125100] | 82298 (24113.99) [72201 to 136900]

8. Secondary Outcome: Urine Concentration of NAG Preoperatively in Recipients
Description: Urine concentration of N-acetyl-D-glucosaminidase (NAG) before the operation
Time Frame: before operation
Population: Urine could not be obtained from the other 46 patients because of anuria.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 8 | 1 | 5
U/L | 20.79 (13.68) | 15.25 (0) | 16.09 (20.71)

9. Secondary Outcome: Urine Concentration of NAG Postoperatively in Recipients
Description: Urine concentration of N-acetyl-D-glucosaminidase (NAG) 1hour, 4hours and 24hours after the artery unclamping in the recipients
Time Frame: within the first 24hours after the artery unclamping
Population: All patients completed the trial and no dropout occured.
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
U/L
  1hour after the artery unclamping | 16.58 (26.94) [4.67 to 54.75] | 18.54 (29.58) [2.99 to 24.02] | 17.06 (31.30) [2.25 to 36.54]
  4hours after the artery unclamping | 3.74 (3.27) [1.3 to 7.12] | 4.45 (10.37) [1.99 to 10.38] | 6.46 (6.92) [1.99 to 13.10]
  24hours after the artery unclamping | 3.73 (7.36) [1.66 to 6.72] | 2.65 (3.01) [1.99 to 5.50] | 4.13 (2.87) [1.69 to 5.80]

10. Secondary Outcome: Urine Concentration of RBP Preoperatively in the Recipients
Description: Urine concentration of retinol binding protein (RBP) before the operation in the recipients
Time Frame: before the operation
Population: No urine could be obtained from the other 46 patients because of anuria.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 8 | 1 | 5
mg/L | 2.222 (0.315) | 2.168 (0) | 1.964 (0.465)

11. Secondary Outcome: Urine Concentration of RBP Postoperatively in the Recipients
Description: Urine concentration of retinol binding protein (RBP) 1hour, 4hours and 24hours after the artery unclamping in the recipients
Time Frame: within the first 24hours after the artery unclamping
Population: All patients completed the trial and no dropout occured.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
mg/L
  1hour after the artery unclamping | 2.18 (0.44) [1.79 to 2.35] | 1.93 (0.42) [1.69 to 2.45] | 2.05 (0.44) [1.92 to 2.30]
  4hours after the artery unclamping | 2.23 (0.28) [1.82 to 2.35] | 1.94 (0.48) [1.66 to 2.35] | 2.27 (0.56) [1.92 to 2.55]
  24hours after the artery unclamping | 2.05 (0.48) [1.69 to 2.35] | 1.91 (0.43) [1.79 to 2.17] | 1.94 (0.50) [1.79 to 2.41]

12. Secondary Outcome: Plasma Concentration of SOD in the Recipients
Description: Plasma concentration of superoxide dismutase (SOD) before the operation, 1hour, 4hours and 24hours after the artery unclamping in the recipients
Time Frame: within 24hours after the operation
Population: All patients completed the trial and no dropout occured.
Measure: Median (Inter-Quartile Range); unit: U/ml
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
U/ml
  before operation | 105.04 (27.08) [77.79 to 121.90] | 96.77 (29.79) [82.91 to 136.46] | 113.51 (23.86) [93.79 to 136.71]
  1hour after the artery unclamping | 88.86 (21.41) [79.19 to 110.06] | 94.90 (28.96) [78.03 to 128.18] | 112.25 (23.92) [91.63 to 115.24]
  4hours after the artery unclamping | 76.47 (28.81) [47.86 to 96.41] | 90.67 (32.49) [69.43 to 115.08] | 89.36 (22.47) [80.01 to 102.75]
  24hours after the artery unclamping | 41.47 (33.83) [33.77 to 95.03] | 64.13 (34.99) [32.92 to 83.01] | 68.04 (29.27) [42.40 to 80.09]

13. Secondary Outcome: Plasma Concentration of MDA in the Recipients
Description: Plasma concentration of malondialdehyde (MDA) before the operation, 1hour, 4hours and 24hours after the artery unclamping in the recipients
Time Frame: within the first 24hours after the operation
Population: All patients completed the trial and no dropout occured.
Measure: Median (Inter-Quartile Range); unit: nmol/ml
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Number analyzed (Participants) | 20 | 20 | 20
nmol/ml
  before operation | 2.96 (0.72) [2.52 to 3.75] | 3.34 (0.70) [2.82 to 3.82] | 3.14 (0.65) [2.91 to 3.66]
  1hour after the artery unclamping | 3.58 (0.80) [3.20 to 4.30] | 4.15 (0.59) [3.51 to 4.63] | 3.91 (0.77) [3.56 to 4.29]
  4hours after the artery unclamping | 3.60 (0.80) [2.90 to 4.21] | 3.46 (0.92) [3.12 to 4.36] | 3.54 (0.84) [3.25 to 4.22]
  24hours after the artery unclamping | 2.97 (0.88) [2.65 to 3.62] | 3.57 (0.72) [2.86 to 3.93] | 3.36 (0.83) [2.87 to 3.86]

ADVERSE EVENTS:
Arm/Group | Control | Donor + RIPC | Recipient +RIPC
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
The trial was conducted only in our hospital and had a relatively small sample size because of the scarcity of relative living donor renal transplantation compared to other surgeries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes